CLINICAL TRIAL: NCT01857089
Title: Characterization of Sitting Postures in Healthy Subjects
Acronym: CaPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CaPAS-DCIC-1204
Record Dates: First submitted 2013-02-01; First posted 2013-05-20 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer; prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pressure Measurement (Experimental)
  Interventions: Device: Orthotest CE

INTERVENTIONS:
Device: Orthotest CE — Orthotest CE is a rigid base mapping system composed by 1024 pressure transducers uniformly distributed in a 35x35 cm surface.
  Orthotest CE is a product manufactured by Vista-Medical. The patient sit on the rigid base during 2 hours to record the pressure and all the data needed for the pilot study.
  Pressure measurement
  Other Names: Orthotest CE mark; Vista-Medical; Mapping system

SUMMARY:
The aim of this study is to assess the intra and inter-subjects variability of the pressure measurement cartography in healthy and well and able volunteers, sitting on a rigid base during two hours.

DETAILED DESCRIPTION:
* The purpose of this study is to understand the formation of pressure sore, to improve the care of paraplegic patients.
* This pilot study is going to help to establish a model in healthy volunteers in the prevention of pressure sores.

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old
* age between 20 and 30 years old
* affiliation to social security or similarly regime

Exclusion Criteria:

* Person with pacemaker
* Person with a history of lumbar pain, chest or/and cervical pain.
* Person with an history of lumbar, chest or/and cervical muscular disorders,
* Person with history of circulatory problems,
* Person with history of skin pathologies at the seat area,
* Protected person referred to in Articles L1121-5 to L1121-8 of the Code of Public Health
* Person having a total annual compensation for the participation in biomedical research higher than €4460.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Assessment of intra and inter-subjects variability of the pressure measurements for the whole population included. | 2 hours
  Sit pressure measurements of all subjects of the study

SECONDARY OUTCOMES:
Correlation between interface pressure measurements and postural data. | 2 hours
  * Sit pressure measurements
  * Video recording

OTHER OUTCOMES:
Correlation between interface pressure measurements and the response to micro electrical stimulation of the buttock. | 2 hours
  * Sit pressure measurements
  * Body composition: body fat mass, lean body mass, water body, bone mineral content etc.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre MOREAU-GAUDRY, MD,PhD, Principal Investigator — INSERM-CIC-IT
Locations (1):
- CIC-IT GrenobleUniversityHospital, Grenoble, France

REFERENCES:
- See also: Related Info — http://www.cic-it-grenoble.fr/